CLINICAL TRIAL: NCT01856790
Title: Effect of Liraglutide on Automated Closed-loop Glucose Control in Type 1 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jennifer Sherr (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Yale University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Sherr, Instructor, Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1211011156
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed Loop Insulin Delivery (Experimental): Each participant recruited into the study will undergo two inpatient closed loop admissions.
  The first admission will be utilizing closed loop control alone, using the Medtronic external Physiological Insulin Delivery (ePID) algorithm. The ePID controller uses a proportional-integral-derivative algorithm modified to include insulin feedback.
  Following the first closed loop admission, each participant is initiated on adjunctive once daily liraglutide therapy. They undergo a 3-4 week dose titration period.
  Participants are then admitted for a second closed loop admission to assess the combined effects of closed loop control with adjunctive once daily liraglutide therapy.
  Interventions: Device: ePID closed loop system; Drug: liraglutide

INTERVENTIONS:
Device: ePID closed loop system — Insulin pump controlled by closed loop unit and algorithm
Drug: liraglutide — Liraglutide is a long-acting analog of human glucagon like peptide-1 (GLP-1) that works as a GLP-1 receptor agonist
  Other Names: Victoza

SUMMARY:
"Closed loop artificial pancreas" systems have been under development for the control of blood sugars in those living with diabetes. These systems consist of a continuous glucose sensor, which sends a signal to a computer program that automatically determines how much insulin to give. The computer program then tells an insulin pump to deliver the insulin. While such systems have been tested under a number of conditions, post-meal blood sugars are difficult to control. This study is designed to see if liraglutide, a glucagon like peptide receptor agonist, can help minimize the post meal blood sugar spikes in subjects with type 1 diabetes while they are on a closed loop system.

DETAILED DESCRIPTION:
Open-label, crossover study comparing the peak post-prandial glucose levels and the incremental post-prandial glucose area under the curve (AUC) during closed loop (CL) control alone and during CL control with liraglutide in an inpatient research setting. Data generated during outpatient baseline evaluation and liraglutide dose titration phases of the study will be compared to assess the short-term efficacy of this agent during open-loop continuous subcutaneous insulin infusion (CSII) pump treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-40 years
2. clinical diagnosis of Type 1 diabetes (T1D) (formal antibody and/or genetic testing will not be required)
3. duration of T1D ≥ 1 year
4. HbA1c ≤ 9 %
5. Treated with CSII for at least 3 months
6. Body weight > 50 kg (to accommodate phlebotomy)
7. Be in good general health without other medical or psychiatric illnesses that would, in the judgment of the investigator, interfere with subject safety or study conduct

Exclusion Criteria:

1. Insulin resistant (defined as requiring > 1.5 units/kg/day at time of study enrollment)
2. Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
3. Use of any medications (besides insulin) known to blood glucose levels, including oral or other systemic glucocorticoid therapy. Inhaled, intranasal, or rectal corticosteroid use is allowed along as not given within 4 weeks of admission to the hospital research unit (HRU). Use of topical glucocorticoids is allowable as long as affected skin area does not overlap with study device sites. Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
4. History of hypoglycemic seizure within last 3 months
5. Anemic (low hematocrit), evidence of renal insufficiency (elevated serum creatinine, BUN) or elevated liver function tests.
6. Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy
7. History of celiac disease gastroparesis, gastroesophageal reflux disease (GERD), disorder of gastric emptying, or disorder of intestinal motility
8. Taking a medication known to affect gastric motility
9. History of pancreatitis, gallstones, alcoholism or high triglyceride levels
10. Personal or family history of thyroid cancer or multiple endocrine neoplasia type 2 (MEN2)
11. Subjects unable to give consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sherr, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Each participant recruited into the study will undergo two inpatient closed loop admissions.
  The first admission will be utilizing closed loop control alone, using the Medtronic external Physiological Insulin Delivery (ePID) algorithm. The ePID controller uses a proportional-integral-derivative algorithm modified to include insulin feedback.
  Following the first closed loop admission, each participant is initiated on adjunctive once daily liraglutide therapy. They undergo a 3-4 week dose titration period.
  Participants are then admitted for a second closed loop admission to assess the combined effects of closed loop control with adjunctive once daily liraglutide therapy.
Period: Closed Loop Control
Arm/Group | All Study Participants
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Closed Loop Control + Liraglutide
Arm/Group | All Study Participants
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Baseline Subject Characteristics: Each participant recruited into the study will undergo two inpatient closed loop admissions.
  The first admission will be utilizing closed loop control alone, using the Medtronic external Physiological Insulin Delivery (ePID) algorithm. The ePID controller uses a proportional-integral-derivative algorithm modified to include insulin feedback.
  Following the first closed loop admission, each participant is initiated on adjunctive once daily liraglutide therapy. They undergo a 3-4 week dose titration period.
  Participants are then admitted for a second closed loop admission to assess the combined effects of closed loop control with adjunctive once daily liraglutide therapy.
Arm/Group | Baseline Subject Characteristics
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Post-prandial Venous Glucose Levels
Description: peak post-prandial venous glucose levels obtained after breakfast, lunch, and dinner between closed loop (CL) alone and CL + liraglutide
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Closed Loop Insulin Delivery: Each participant recruited into the study will undergo two inpatient closed loop admissions.
  The first admission will be utilizing closed loop control alone, using the Medtronic external Physiological Insulin Delivery (ePID) algorithm. The ePID controller uses a proportional-integral-derivative algorithm modified to include insulin feedback.
- Closed Loop + Liraglutide: Following the first closed loop admission, each participant is initiated on adjunctive once daily liraglutide therapy. They undergo a 3-4 week dose titration period.
  Participants are then admitted for a second closed loop admission to assess the combined effects of closed loop control with adjunctive once daily liraglutide therapy.
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
mg/dL | 98 (24) | 76 (17)
Statistical Analysis 1: Comparison: Closed Loop Insulin Delivery vs Closed Loop + Liraglutide; Test type: Superiority or Other; p = 0.05, Wilcoxon Matched Pairs signed rank tests

2. Secondary Outcome: the Incremental Meal-related Glucose Area Under Curve (AUC)
Time Frame: 5-hour post prandial period after breakfast, lunch, and dinner
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
mg*hr/dL | 789 (176) | 500 (151)
Statistical Analysis 1: Comparison: Closed Loop Insulin Delivery vs Closed Loop + Liraglutide; Test type: Superiority or Other; p = 0.002, Wilcoxon Matched Pairs signed rank tests

3. Other Pre Specified Outcome: Mean 24-hour Glucose Levels
Time Frame: 24- hours
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Closed Loop Insulin Delivery; Closed Loop + Liraglutide: Following the first closed loop admission, each participant is initiated on adjunctive once daily liraglutide therapy. They undergo a 3-4 week dose titration period.
  Participants are then admitted for a second closed loop admission to assess the combined effects of closed loop control with adjunctive once daily liraglutide therapy.
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
mg/dL | 130 (51) | 135 (45)

4. Other Pre Specified Outcome: Mean Time to Peak Post-meal Glucose Value
Time Frame: 5- hour postprandial period
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
hours | 1.8 (0.5) | 1.8 (0.6)
Statistical Analysis 1: Comparison: Closed Loop Insulin Delivery vs Closed Loop + Liraglutide; Test type: Superiority or Other; p = 0.97, Wilcoxon Matched Pairs signed rank tests

5. Other Pre Specified Outcome: Mean Daytime Glucose Levels
Time Frame: 8a.m.-11p.m.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- ePID Closed Loop System Without Liraglutide: ePID closed loop system alone
  ePID closed loop system: Insulin pump controlled by closed loop unit and algorithm
- ePID Closed Loop System With Liraglutide: liraglutide + ePID closed loop system
  ePID closed loop system: Insulin pump controlled by closed loop unit and algorithm
  liraglutide: Liraglutide is a long-acting analog of human glucagon-like peptide 1 (GLP-1) that works as a GLP-1 receptor agonist
Arm/Group | ePID Closed Loop System Without Liraglutide | ePID Closed Loop System With Liraglutide
Number analyzed (Participants) | 11 | 11
mg/dL | 143 (55) | 146 (47)

6. Other Pre Specified Outcome: Incremental Glucagon Peak
Time Frame: 5 hours
Measure: Mean (Standard Deviation); unit: pg/mL/min
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 10 | 10
pg/mL/min | 29 (16) | 35 (20)

7. Other Pre Specified Outcome: AUC Plasma Glucagon During MMTT
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 10 | 10
pg*min/mL | 1904 (651) | 1801 (906)

8. Other Pre Specified Outcome: Differences in Daily Insulin Requirements
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units
Groups:
- Pre-Liraglutide Treatment: Baseline characteristics prior to liraglutide therapy
- Post-Liraglutide Treatment: Characteristics following 3 week outpatient dose titration phase of liraglutide
Arm/Group | Pre-Liraglutide Treatment | Post-Liraglutide Treatment
Number analyzed (Participants) | 11 | 11
units | 51.5 (14) | 37.5 (12.9)
Statistical Analysis 1: Comparison: Pre-Liraglutide Treatment vs Post-Liraglutide Treatment; Test type: Superiority or Other; p = .001, Wilcoxon Matched Pairs signed rank tests

9. Other Pre Specified Outcome: Prandial Insulin Delivery During Closed Loop Therapy
Time Frame: Average of the 5-hour post prandial period for breakfast, lunch, dinner combined
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
units | 22.6 (8.4) | 16.3 (8.3)
Statistical Analysis 1: Comparison: Closed Loop Insulin Delivery vs Closed Loop + Liraglutide; Test type: Superiority or Other; p = 0.005, Wilcoxon Matched Pairs signed rank tests

10. Other Pre Specified Outcome: Mean Nocturnal Glucose Levels
Time Frame: 11p.m.-6a.m.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Insulin Delivery | Closed Loop + Liraglutide
Number analyzed (Participants) | 11 | 11
mg/dL | 104 (23) | 113 (24)

ADVERSE EVENTS:
Description: Adverse events were recorded in categories with gastrointestinal disorders encompassing nausea, decreased appetite, constipation, bloating and/or diarrhea
Groups:
- Closed Loop Only: Each participant recruited into the study will undergo two inpatient closed loop admissions.
  The first admission will be utilizing closed loop control alone, using the Medtronic external Physiological Insulin Delivery (ePID) algorithm. The ePID controller uses a proportional-integral-derivative algorithm modified to include insulin feedback
Arm/Group | Closed Loop Only | Closed Loop + Liraglutide
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Only (N=13) | Closed Loop + Liraglutide (N=11)
gastrointestinal distress (Gastrointestinal disorders) | 0 (0) | 6 — nausea, decreased appetite, constipation, bloating, and/or diarrhea
headache (Nervous system disorders) | 0 | 6 — headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No